CLINICAL TRIAL: NCT04674917
Title: Effects of Decompression on Pain, Range of Motion and Function in Patient With Acute vs Chronic Lumbar Radiculopathy
Brief Title: Effects of Decompression in Patient With Acute vs Chronic Lumbar Radiculopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/LHR/20/1051 Mariam Waseem
Record Dates: First submitted 2020-12-16; First posted 2020-12-19 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Lumbar Radiculopathy
Keywords: Decompression, radiculopathy, acute, chronic
MeSH Terms: conditions — Radiculopathy; Bronchiolitis Obliterans Syndrome | interventions — Decompression; Transcutaneous Electric Nerve Stimulation; Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Decompression + Hot pack, TENS, Mobilization, Exercise Therapy
  Interventions: Other: Decompression + Hot pack, TENS, Mobilization, Exercise Therapy
- Group B (Experimental): Decompression + Hot pack, TENS, Mobilization, Exercise Therapy
  Interventions: Other: Decompression + Hot pack , TENS , Mobilization , Exercise Therapy
- Group C (Other): Hot pack , TENS, Mobilization, Exercise therapy
  Interventions: Other: Hot pack , TENS, Mobilization, Exercise therapy

INTERVENTIONS:
Other: Decompression + Hot pack, TENS, Mobilization, Exercise Therapy — Group A which includes the acute group to study the effects of decompression we will apply the three main basic treatments along with decompression which is our main goal..
  The basic treatments are
  1. Hot Pack
  2. TENSE
  3. Mobilization ( on lumbar L1 toL5 ) Our first modality which is hot pack will be given to the patients for a duration of 15 minutes The next modality TENSE will be given for 10 minutes
  The third treatment which is mobilization will be given 1 time on each joint of lumbar spine All these treatments must given in combination with the decompression.
  Arms: Group A
Other: Decompression + Hot pack , TENS , Mobilization , Exercise Therapy — Group B which includes the chronic group to study the effects of decompression we will apply the three main basic treatments along with decompression which is our main goal..
  The basic treatments are
  1. Hot Pack
  2. TENSE
  3. Mobilization ( on lumbar L1 toL5 )
  Our first modality which is hot pack will be given to the patients for a duration of 15 minutes The next modality TENSE will be given for 10 minutes
  The third treatment which is mobilization will be given 1 time on each joint of lumbar spine All these treatments must given in combination with the decompression.
  Arms: Group B
Other: Hot pack , TENS, Mobilization, Exercise therapy — Group C which is our control group to compare it with the groups A and B to study the effects of decompression on lumbar radiculopathy The basic treatments are
  1. Hot Pack
  2. TENSE
  3. Mobilization ( on lumbar L1 toL5 )
  Our first modality which is hot pack will be given to the patients for a duration of 15 minutes The next modality TENSE will be given for 10 minutes
  The third treatment which is mobilization will be given 1 time on each joint of lumbar spine It is kept in mind that in this group we will not apply the decompression along with the above treatments.
  Arms: Group C

SUMMARY:
The study will be done to evaluate the effectiveness of Lumbar Spinal Decompression in patients with acute vs chronic lumbar radiculopathy. Study design will be Randomized control trial and sample size will be 30. Duration of study was of 6 month, convenient sampling was done. Data will be collected from DHQ Daska were randomly allocated in three groups via lottery method, baseline assessment was done. Patients of both gender (male and female) from 18 to 50 years with lumbar radiculopathy diagnosed through X-ray and physical examination will be included. Patients with systemic soft tissue and bony diseases will be excluded. Intervention duration of 4 weeks, 3 sessions in a week. Decompression of lumbar spine will be given once in a week. Whole procedure of treatment program will given to patients and written informed consent will be taken. Basic tools will be Visual analog scale (VAS), SLR, ODI, Inclinometer. Data was analyzed by using SPSS version 21

DETAILED DESCRIPTION:
Low back pain (LBP) is one of the most common musculoskeletal conditions treated by physical therapists. Although lumbar traction is frequently used by physical therapists in the treatment of patients with LBP. We will use Manual Lumber Spinal Traction on patients with acute vs chronic lumber radiculopathy. The current study will determine the effect of decompression in relieving pain, increase range of motion and improving function in patients of acute and chronic lumbar radiculopathy. Lumbar traction (LT) is routinely used on its own or in conjunction with other treatments for the management of lumbar sciatica. We will use Manual lumbar traction along with hot pack, tens, mobilization and exercise therapy. Intervention duration of 4 weeks, 3 sessions in a week. Decompression of lumbar spine will be given once in a week.

ELIGIBILITY:
Inclusion Criteria:

* history of radicular pain with straight leg raise (SLR).
* Patients in the acute phase of (up to 6 weeks) included in group A
* Patients in chronic phase of (more than 6 weeks) included in group B

Exclusion Criteria:

* Any systemic soft tissue and bony disease.
* Patient with spinal tuberculosis, spinal fractures, pregnancy, cancer.
* Any recent surgery.
* Patient with any cervical or thoracic problem.
* Patients with any other serious pathology/red flags

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 4th week
  A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured

SECONDARY OUTCOMES:
MODIFIED OSWESTRY LOW BACK PAIN DISABILITY QUESTIONNAIRE | 4th Week
  The Oswestry Disability Index (also known as the Oswestry Low Back Pain Disability Questionnaire) is an extremely important tool that researchers and disability evaluators use to measure a patient's permanent functional disability. The test is considered the 'gold standard' of low back functional outcome tools

OTHER OUTCOMES:
Inclinometer | 4th Week
  An inclinometer or clinometer is an instrument used for measuring angles of slope (or tilt), elevation, or depression of an object with respect to gravity's direction.

CONTACTS AND LOCATIONS:
Overall Officials: Syed Shakil Ur Rehman, Principal Investigator — Riphah International University
Locations (1):
- DHQ hospital, Daska Kalan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheng YH, Hsu CY, Lin YN. The effect of mechanical traction on low back pain in patients with herniated intervertebral disks: a systemic review and meta-analysis. Clin Rehabil. 2020 Jan;34(1):13-22. doi: 10.1177/0269215519872528. Epub 2019 Aug 28. PMID 31456418
- [Background] Swanson BT, Riley SP, Cote MP, Leger RR, Moss IL, Carlos J Jr. Manual unloading of the lumbar spine: can it identify immediate responders to mechanical traction in a low back pain population? A study of reliability and criterion referenced predictive validity. J Man Manip Ther. 2016 May;24(2):53-61. doi: 10.1179/2042618614Y.0000000072. PMID 27559274
- [Background] Rubinic DM, Koo V, Dudley J, Owens SC. Changes in Spinal Height After Manual Axial Traction or Side Lying: A Clinical Measure of Intervertebral Disc Hydration Using Stadiometry. J Manipulative Physiol Ther. 2019 Mar-Apr;42(3):187-194. doi: 10.1016/j.jmpt.2019.03.005. Epub 2019 May 9. PMID 31078315
- [Background] Asiri F, Tedla JS, D Alshahrani MS, Ahmed I, Reddy RS, Gular K. Effects of patient-specific three-dimensional lumbar traction on pain and functional disability in patients with lumbar intervertebral disc prolapse. Niger J Clin Pract. 2020 Apr;23(4):498-502. doi: 10.4103/njcp.njcp_285_19. PMID 32246656
- [Background] Mo Z, Li D, Zhang R, Chang M, Yang B, Tang S. Comparisons of the Effectiveness and Safety of Tuina, Acupuncture, Traction, and Chinese Herbs for Lumbar Disc Herniation: A Systematic Review and Network Meta-Analysis. Evid Based Complement Alternat Med. 2019 Mar 20;2019:6821310. doi: 10.1155/2019/6821310. eCollection 2019. PMID 31015852
- [Background] Mitchell UH, Beattie PF, Bowden J, Larson R, Wang H. Age-related differences in the response of the L5-S1 intervertebral disc to spinal traction. Musculoskelet Sci Pract. 2017 Oct;31:1-8. doi: 10.1016/j.msksp.2017.06.004. Epub 2017 Jun 9. PMID 28624722
- [Background] Isner-Horobeti ME, Dufour SP, Schaeffer M, Sauleau E, Vautravers P, Lecocq J, Dupeyron A. High-Force Versus Low-Force Lumbar Traction in Acute Lumbar Sciatica Due to Disc Herniation: A Preliminary Randomized Trial. J Manipulative Physiol Ther. 2016 Nov-Dec;39(9):645-654. doi: 10.1016/j.jmpt.2016.09.006. Epub 2016 Nov 9. PMID 27838140
- [Background] Tadano S, Tanabe H, Arai S, Fujino K, Doi T, Akai M. Lumbar mechanical traction: a biomechanical assessment of change at the lumbar spine. BMC Musculoskelet Disord. 2019 Apr 9;20(1):155. doi: 10.1186/s12891-019-2545-9. PMID 30961554
- [Background] Creighton D, Schweiger A, Cubr S. Immediate Effects of Side Lying Manual Lumbar Traction in Patients with Painful Active Lumbar Motion. Journal of International Academy of Physical Therapy Research. 2017;8(1):1071-6.
- [Background] Oh H, Choi S, Lee S, Choi J, Lee K. The impact of manual spinal traction therapy on the pain and Oswestry disability index of patients with chronic back pain. J Phys Ther Sci. 2018 Dec;30(12):1455-1457. doi: 10.1589/jpts.30.1455. Epub 2018 Nov 21. PMID 30568333
- [Background] Kisner C, Colby LA, Borstad J. Therapeutic exercise: foundations and techniques: Fa Davis; 2017.
- [Background] Thackeray A, Fritz JM, Childs JD, Brennan GP. The Effectiveness of Mechanical Traction Among Subgroups of Patients With Low Back Pain and Leg Pain: A Randomized Trial. J Orthop Sports Phys Ther. 2016 Mar;46(3):144-54. doi: 10.2519/jospt.2016.6238. Epub 2016 Jan 26. PMID 26813755
- [Background] Szulc P, Wendt M, Waszak M, Tomczak M, Cieslik K, Trzaska T. Impact of McKenzie Method Therapy Enriched by Muscular Energy Techniques on Subjective and Objective Parameters Related to Spine Function in Patients with Chronic Low Back Pain. Med Sci Monit. 2015 Sep 29;21:2918-32. doi: 10.12659/MSM.894261. PMID 26418868
- [Background] Lo WLA, Lei D, Leng Y, Huang H, Wang B, Yu Q, Li L. Impact of nonsurgical spinal decompression on paraspinal muscle morphology and mechanical properties in young adults with low back pain. J Int Med Res. 2020 Jul;48(7):300060520919232. doi: 10.1177/0300060520919232. PMID 32723102
- [Background] Hallur SS, Brismee JM, Sizer PS, Dierick F, Dewan BM, Thiry P, Sobczak S. Three-Dimensional Spinal Position With and Without Manual Distraction Load Increases Spinal Height. J Manipulative Physiol Ther. 2020 May;43(4):267-275. doi: 10.1016/j.jmpt.2019.04.007. Epub 2020 Jul 21. PMID 32709513